CLINICAL TRIAL: NCT02220231
Title: Echocardiographic Evaluation of the Change on Pulmonary Blood Flow and Cardiac Function Induced by Capnothorax During One Lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 4-2014-0492
Record Dates: First submitted 2014-08-06; First posted 2014-08-19 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Mediastinal Tumors
Keywords: mediastinal mass, one-lung ventilation, capnothorax, transesophageal echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- capnothorax group (Experimental): After patient positioning, the capnothorax will be created by insufflation of carbon dioxide in patients undergoing video-assisted thoracoscopic extended thymectomy.
  Interventions: Procedure: capnothorax

INTERVENTIONS:
Procedure: capnothorax — After patient positioning, the capnothorax will be created by insufflation of carbon dioxide in patients undergoing video-assisted thoracoscopic extended thymectomy.
  Other Names: VATET, capnothorax, TEE

SUMMARY:
Video-assisted thoracoscopic extended thymectomy (VATET) is a minimally-invasive method for excision of mediastinal mass instead of open thymectomy. The iatrogenic capnothorax with one-lung ventilation during VATET may cause hemodynamic instability due to the compression of intrathoracic structures. The purpose of this study is to evaluate the effects of capnothorax on the pulmonary blood flow and cardiac function during the VATET by using the transesophageal echocardiography.

DETAILED DESCRIPTION:
Video-assisted thoracoscopic extended thymectomy (VATET) is a minimally-invasive method for excision of mediastinal mass instead of open thymectomy. The iatrogenic capnothorax with one-lung ventilation during VATET may cause hemodynamic instability due to the compression of intrathoracic structures. The purpose of this study is to evaluate the effects of capnothorax on the pulmonary blood flow and cardiac function during the VATET by using the transesophageal echocardiography

ELIGIBILITY:
Inclusion Criteria:

1. Above 20 years of age.
2. American Society of Anesthesiologists (ASA) Physical Status I, II, III.
3. Thoracic surgical procedure (video-assisted thoracoscopic extended thymectomy )

Exclusion Criteria:

1. Severe functional liver or kidney disease
2. Diagnosed HF ( NYHA class >3)
3. Arrhythmia or received treatment with antiarrhythmic drug .
4. Exceed BMI > 30 kg/ m2
5. COPD
6. Pathologic esophageal lesion (esophageal stricture or varix )
7. Pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The changes of the echocardiographic indices | four time points during the operation. (1)10 min after induction (baseline); (2) 1 min after CO2 insufflation; (3)10 min after of CO2 insufflation; and (4)20 min after CO2 insufflation
  pulmonary blood flow = PVA(cross sectional area of LUPV) x VTI(velocity time integral) x HR , Fractional area change = [(LVAd-LVAs)/LVAd] × 100 Ejection fraction = [(LVEDV(LV end-diastolic volume) -LVESV(LV end-systolic volume)/LVEDV] × 100

SECONDARY OUTCOMES:
The changes of the oxygenation and respiratory dynamic parameters | four time points during the operation, an expected average of 3 hours. (1)10 min after induction (baseline); (2) 1 min after CO2 insufflation; (3)10 min after of CO2 insufflation; and (4)20 min after CO2 insufflation
  shunt fraction Qs/Qt = (CcO2- CaO2)/(CcO2- CvO2) CcO2 = Hgb x 1.34 x ScO2 + PcO2 x 0.003, lung compliance : Compliance= Vt / Pplat, physiologic dead space : Vd/Vt = 1.14 x (PaCO2 - PETCO2)/PaCO2- 0.005